CLINICAL TRIAL: NCT00642122
Title: A Randomized, Blinded, Multicenter, Parallel Study Comparing the Efficacy and Safety of Pulmicort Respules at 0.5mg QD, 1.0mg QD, 1.0mg Bid, 2.0mg Bid and Pulmicort Turbuhaler at 4.00mcg Bid on Adolescents (12 Yrs of Age and Older) With Adults With Moderate to Severe Asthma.
Brief Title: Adults With Moderate to Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SD-004-0764; D5257L00012
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort; budesonide; respules; turbuhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pulmicort RESPULES
  Interventions: Drug: Budesonide
- 2 (Experimental): Pulmicort TURBUHALER
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — 0.5mg once daily
  Other Names: Pulmicort RESPULES
  Arms: 1
Drug: Budesonide — 1mg once daily
  Other Names: Pulmicort RESPULES
  Arms: 1
Drug: Budesonide — 1mg twice daily
  Other Names: Pulmicort RESPULES
  Arms: 1
Drug: Budesonide — 2mg once daily
  Other Names: Pulmicort RESPULES
  Arms: 1
Drug: Budesonide — 4.00mcg twice daily
  Other Names: Pulmicort TURBUHALER
  Arms: 2

SUMMARY:
A study to compare the safety and effectiveness of 5 different ways of taking Pulmicort when given to asthma patients aged 12 years and above.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 12 or over who have asthma
* Ability to properly use an electronic diary
* Able and willing to nebulize for up to 20 minutes every morning and evening

Exclusion Criteria:

* Hospitalised at least one once or required emergency treatment due to asthma in the previous 6 months
* Planned hospitalisation during the study
* pregnant women or women planning to become pregnant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second in patients allocated treatment with Pulmicort REPSULES at 0.5mg and 2.0mg. | Day -14, 1, and every 28 days thereafter

SECONDARY OUTCOMES:
Percentage of symptom free days | Day -14, 1, and every 28 days thereafter
Percentage of symptom free nights | Day -14, 1, and every 28 days thereafter
Percentage of symptom free 24-hours | Day -14, 1, and every 28 days thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Andersson, Study Director — AstraZeneca